CLINICAL TRIAL: NCT05781477
Title: Effect of Breastfeeding Training Program and Nurse-led Breastfeeding Online Counselling System (BMUM) for Mothers: Randomized Controlled Study
Brief Title: Effect of Breastfeeding Training Program and System (BMUM) for Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Şahika ŞİMŞEK ÇETİNKAYA, PhD,Dr., Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-6/16.06.2020
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bmum GROUP (Experimental): Mothers in this group were given supportive breastfeeding support with web based
  Interventions: Behavioral: Bmum supportive system
- control group (No Intervention): Mothers in the control and intervention groups were given standard care based on the Baby-Friendly Hospital Intervention Standard.

INTERVENTIONS:
Behavioral: Bmum supportive system — Bmum is a web-based online tracking system that aims to improve positive attitude about breastfeeding
  Arms: Bmum GROUP

SUMMARY:
The goal of the study was to investigate effect of breastfeeding training program and nurse-led breastfeeding online counselling system (BMUM) on mothers' breastfeeding self-efficacy, breastfeeding attitudes, breastfeeding problems and postpartum depression we hypothesized that there would be differences between BG and CG groups in terms of breastfeeding self-efficacy, breastfeeding problems, postpartum depression and breastfeeding frequency. This was a randomized controlled trial. Participants were randomly assigned to the breastfeeding group (BG; n = 36), or control group (CG; n = 36). Control group will receive only standart care breastfeeding group will receive standart care and web based breastfeeding support. Breastfeeding attitudes, infant feeding attitude breastfeeding problems and postpartum depression will assessment. The assesment point will be 32-37 gestational week, postpartum 1st day, 1st week, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old,
* Primipara with a singleton pregnancy
* 32- and 37-weeks of gestation,
* Willingness to participate in the workshop program

Exclusion Criteria:

* Having a chronic illness
* Having pre-term labor or an abnormal fetal screening
* Had a psychiatric disorder or anxiety disorder
* Having any other high-risk complications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self efficacy change on five points between groups | 32-37 weeks 1st. day 1. week 3rd months 6th months
  Breastfeeding Self efficacy short form scale will use to assessment breasfeeding self efficacy. Total scores vary from 14 to 70, with higher scores indicating greater self-efficacy
Infant feeding attitude change on five points between groups | 32-37 weeks 1st. day 1. week 3rd months 6th months
  Iowa Infant Feeding Attitude Scale (IIFAS) will use to assessment infant feeding attitude Higher scores indicate a more favorable attitude toward newborn feeding
Postpartum depression change on four points between groups. | 1st. day 1st. week 3rd months 6th months
  Edinburgh Postnatal Depression Scale (EPDS) will use to assesment postpartum depression. The total score ranges from 0 to 30, with higher scores suggesting a higher level of depression symptoms.
breast problems between two groups on 1 st week | 1st week
  breast problem will assesment with breastfeeding problems questionnaire. number and percent will use to evaluate.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kastamonu University, Merkez, Kastamonu
  - Şahika Şimşek Çetinkaya, Merkez, Kastamonu